CLINICAL TRIAL: NCT07307690
Title: Comparison of the Effectiveness of 8-week vs 12-week Physical Exercise Programmes in Patients With Colorectal Cancer
Brief Title: 8 Weeks vs 12 Weeks Physical Exercise Programmes in Colorectal Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, CARLOS MARTIN SANCHEZ, PhD, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ComparisonCCRDic2025
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Oncology; Chemotherapy-Induced Peripheral Neuropathy
Keywords: Exercise; Cancer; Colorectal cancer; wellbeing; Mental health
MeSH Terms: conditions — Neoplasms; Motor Activity; Colorectal Neoplasms; Psychological Well-Being | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The investigators propose a 8 vs 12-week intervention with therapeutic strength exercise in patients with colorectal cancer who are receiving chemotherapy treatment.
  Interventions: Other: Exercise; Other: Physical activity recommendations
- Control group (Experimental): They will be provided with clear and concrete recommendations of activities for the user to perform the rest of the days of the week in order to increase their level of physical activity and increase weekly metabolic expenditure.
  Interventions: Other: Physical activity recommendations

INTERVENTIONS:
Other: Exercise — There will be 2 weekly sessions of 50 minutes, always guided by a physiotherapist, with the following distribution:
  1.- Warm-up: 15 minutes of global exercises of strength and resistance, focusing on the areas that are going to be worked as a priority in that session.
  Strength training: 6 to 8 strength exercises of large muscle groups. The approximate duration will be 25 minutes.
  3.- Cool down / cool down: Combination of breathing exercises and stretching, 10 minutes.
  Monitoring with activity bracelets.
  Arms: Exercise group
Other: Physical activity recommendations — They will be provided with a physical activity plan to be followed on a weekly basis.

SUMMARY:
Chemotherapy is a cornerstone in the treatment of colon cancer; however, its effects extend beyond malignant cells. Because chemotherapeutic agents target rapidly dividing cells, they can also damage healthy tissues, resulting in a range of adverse effects. Among the most prevalent is peripheral neuropathy, a disorder of the peripheral nervous system characterized by symptoms such as tingling, numbness, pain, and weakness in the extremities.

Chemotherapy-induced peripheral neuropathy poses a significant challenge for patients with colon cancer, as it further compromises quality of life during an already demanding phase of treatment. Damage to sensory and motor nerves interferes with the ability to perform daily activities and diminishes physical capacity, thereby intensifying both the physical and psychological burden associated with the disease.

Nevertheless, certain interventions may help mitigate these negative effects, with physical exercise emerging as a particularly promising strategy. Although it may appear counterintuitive, regular physical activity has been shown to exert beneficial effects on peripheral neuropathy. Exercise enhances blood circulation, supports the regeneration of damaged peripheral nerves, and helps reduce neuropathic pain and discomfort, ultimately improving functional performance.

It is important to emphasize that exercise interventions should be individually tailored and conducted under appropriate medical supervision. Consequently, the integration of chemotherapy with a carefully designed exercise program represents a comprehensive approach to managing both the disease and its treatment-related side effects, contributing to an improved quality of life for patients with colon cancer throughout their recovery process.

DETAILED DESCRIPTION:
1. Introduction Colon cancer is one of the leading causes of morbidity and mortality worldwide, with an increasing incidence in many developed countries. In Spain, it is one of the most common types of cancer, accounting for approximately 15% of all cancer cases diagnosed, with an incidence of around 41,000 new cases annually. The mortality associated with colon cancer is significant, although there have been notable improvements in five-year survival rates, which currently stand at around 65%, thanks to advances in treatments and early diagnosis. Early diagnosis is crucial and has been facilitated by screening programs such as colonoscopy and fecal occult blood tests, which allow the detection of precancerous lesions and early-stage cancer. Treatments for colon cancer include surgery, radiotherapy, immunotherapy, and notably, chemotherapy. Chemotherapy is especially relevant in adjuvant treatment to reduce the risk of postoperative recurrence and in metastatic disease to control tumor growth and prolong survival. Modern chemotherapeutic agents, combined with targeted and supportive therapies, have significantly improved treatment outcomes, providing patients with better recovery prospects and an enhanced quality of life during and after treatment.

Chemotherapy is a crucial treatment in the fight against colon cancer, but unfortunately, its impact is not limited solely to cancer cells. Chemotherapeutic agents, designed to target rapidly growing cells, also affect healthy tissues, leading to various side effects. One of the most common adverse effects is peripheral neuropathy, a condition that affects the peripheral nerves and can manifest as sensations of tingling, numbness, pain, or weakness in the limbs. Chemotherapy-induced peripheral neuropathy can be especially challenging for patients with colon cancer, as it further worsens the quality of life during an already difficult period. The nerves responsible for motor and sensory function are compromised, affecting the patient's ability to perform daily activities and weakening their physical endurance.

This phenomenon adds to the emotional and physical burden of battling cancer. However, there are tools that can positively influence these adverse effects, such as physical exercise. Although it may seem contradictory, regular physical exercise has been shown to have beneficial effects on peripheral neuropathy. Physical exercise can improve blood circulation and promote the regeneration of damaged peripheral nerves.

Additionally, exercise helps alleviate the pain and discomfort associated with neuropathy, thereby strengthening patients' functional capacity.

Scientific research has demonstrated that physical exercise has multiple benefits for cancer patients, beyond alleviating peripheral neuropathy. Various studies have indicated that regular physical activity can significantly improve immune function, which is crucial for patients undergoing treatments that weaken the immune system. Exercise helps increase the production and efficiency of immune cells, enhancing the body's ability to fight infections and potentially inhibiting the growth of cancer cells.

Furthermore, physical exercise has been associated with a reduction in cancer-related fatigue, one of the most debilitating symptoms experienced by patients during and after treatment. Fatigue can severely limit patients' ability to engage in daily activities and reduce their quality of life. Research has shown that structured exercise programs, including aerobic and resistance activities, can diminish the sensation of fatigue and improve energy levels and mood, allowing patients to lead more active and fulfilling lives.

Physical activity also plays a vital role in weight management and body composition, important factors for cancer survival and recovery. Obesity and overweight are associated with poorer prognosis in many types of cancer, including colon cancer. Regular exercise helps maintain a healthy weight, reduce body fat, and improve muscle mass, which not only contributes to a better quality of life but can also reduce the risk of cancer recurrence and improve overall treatment outcomes. Scientific evidence strongly supports the inclusion of physical exercise as an integral part of the treatment plan for cancer patients.

It is essential to highlight that any exercise plan should be tailored to the individual capabilities of each patient, and medical supervision is crucial. Therefore, the combination of chemotherapy and carefully planned physical exercise offers a comprehensive strategy to address both the disease and its side effects, providing colon cancer patients with a better quality of life during their recovery journey.

It is of vital importance to conduct research on the implementation of physical exercise programs in patients with colon cancer to control all the previously mentioned symptoms, such as peripheral neuropathy, fatigue, decreased immune function, and weight management.

These investigations should focus on developing personalized and safe exercise protocols that can be effectively integrated into standard oncological treatment. By generating robust evidence on the benefits and best practices for including physical exercise in the management of colon cancer, patient quality of life can be significantly improved, treatment outcomes optimized, and the incidence of debilitating side effects reduced.

Moreover, these studies can provide crucial data to guide healthcare professionals in prescribing specific exercise programs, ensuring that patients receive evidence-based interventions that maximize their physical and emotional well-being throughout the recovery process.

Therefore, this project sets the following study objectives. As the main objective, this study aims to evaluate and compare the effectiveness of an 8-week versus a 12-week exercise programme in improving chemotherapy-induced peripheral neuropathy in patients with colorectal cancer. And as secondary objectives, the following:

1. To assess the impact of a strength exercise program on quality of life in patients with colorectal cancer undergoing chemotherapy treatment.
2. To evaluate the impact of a strength exercise program on body mass index in patients with colorectal cancer undergoing chemotherapy treatment.
3. To evaluate the impact of a strength exercise program on maximum oxygen consumption in patients with colorectal cancer undergoing chemotherapy treatment.
4. To evaluate the impact of a strength exercise program on anxiety and depression in patients with colorectal cancer undergoing chemotherapy treatment.
5. To evaluate the impact of a strength exercise program on fatigue in patients with colorectal cancer undergoing chemotherapy treatment.
6. To evaluate the impact of a strength exercise program on sleep quality in patients with colorectal cancer undergoing chemotherapy treatment.

Study Design and Setting A double-blind randomized controlled trial was conducted at the Faculty of Nursing and Physiotherapy, University of Salamanca (Spain), following the Consolidated Standards of Reporting Trials (CONSORT) Statement. The current treatment protocol is described according to the recommendations of SPIRIT. The protocol for this trial received approval from the Ethics Committee of the University of Salamanca (record number 1209) and was conducted in accordance with the Declaration of Helsinki. The clinical trial was registered in ClinicalTrials.gov (registration number NCT06404359).

Participants diagnosed with colorectal cancer undergoing adjuvant chemotherapy treatment were recruited from the outpatient clinics of the Day Oncology Hospital at the University Assistance Complex of Salamanca and from the Asociación Española Contra el Cáncer (AECC).

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with colorectal cancer and who are receiving chemotherapy treatment.
* Sedentary people who have not performed physical activity in the last 8 weeks.
* Ability to understand the evaluation tests and the performance of the exercises.
* Presence of XXX symptoms (If we focus on neuropathy, it should be inclusion criteria).
* Voluntary participation in the study.

Exclusion Criteria:

- Present contraindication/s for physical exercise (musculoskeletal diseases, severe cardiovascular disease, bone metastases,...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy-induced neuropathy | Baseline and immediately after the intervention
  The EORTC CIPN20 questionnaire will be used.This questionnaire contains 20 items on which patients rate their experience for each symptom during the previous week using scores from 1 (not at all) to 4 (very much). The sum score was obtained by adding the scores of items 1 to 19 resulting in a sum score range of 19 to 76, which was termed CIPN20 sum1-19.

SECONDARY OUTCOMES:
Wellbeing | Baseline and immediately after the intervention
  It will be evaluated through the the EORTC QLG Core Questionnaire (EORTC QOL-30) quality of life questionnaire in its specific version for colorectal cancer EORT QLQ-CR30. Scores can range from 0 (worst quality of life) to 100 (best quality of life), with higher values indicating better quality of life in the areas evaluated.
Body Mass Index | Baseline and immediately after the intervention
  Obtained from the participant's weight and height.
Mental health | Baseline and immediately after the intervention
  They will be evaluated through the Hospital Anxiety and Depression Scale (HADS). Scores on the HADS can be interpreted as follows:
  Anxiety:
  0-7: Absence of clinically significant anxiety. 8-10: Possible presence of clinically significant anxiety. 11 or more: Clinically significant anxiety.
  Depression:
  0-7: Absence of clinically significant depression. 8-10: Possible presence of clinically significant depression. 11 or more: Clinically significant depression.
Sleep quality | Baseline and immediately after the intervention
  Will be evaluated through the Minimal Insomnia Symptom Scale (MISS). Each question is scored on a scale of 0 to 4, where 0 indicates that the symptom is not present and 4 indicates a very severe presence of the symptom. Therefore, the total score on the MISS can range from 0 to 12 points.
  Interpretations of the MISS scores may be as follows:
  0-3 points: Absence or minimal presence of insomnia symptoms. 4-6 points: Mild insomnia symptoms. 7-9 points: Moderate insomnia symptoms. 10-12 points: Severe insomnia symptoms.

IPD SHARING:
Plan to Share IPD: Undecided
Upon request by e-mail to the principal investigator

REFERENCES:
- [Background] Martin-Sanchez C, Fernandez-Rodriguez EJ, Lopez-Mateos Y, Garcia-Martin A, Fonseca-Sanchez E, Sanchez-Gonzalez JL. Effects of a Resistance Exercise Program in Patients with Colorectal Cancer Undergoing Chemotherapy Treatment: A Randomized Controlled Trial Study Protocol. J Clin Med. 2024 Jul 31;13(15):4478. doi: 10.3390/jcm13154478. PMID 39124745